CLINICAL TRIAL: NCT01635712
Title: A Phase 1, Open-label, Dose-escalation Study of the Safety of SNX-5422 Mesylate in Subjects With Refractory Hematological Malignancies
Brief Title: Safety and Pharmacology Study of SNX-5422 in Subjects With Refractory Hematological Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Esanex Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNX-5422-CLN1-005
Record Dates: First submitted 2012-07-04; First posted 2012-07-09 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Cancer
Keywords: Hematological Malignancy; Hsp90
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms | interventions — SNX-5422

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SNX-5422 (Experimental): Open label administration of SNX-5422 capsules every other day (QOD) for 21 days on a 28 day cycle. Dose escalation will be based on safety outcomes defined as 1 or less dose limiting toxicities during the first 28 day cycle at any dose level
  Interventions: Drug: SNX-5422

INTERVENTIONS:
Drug: SNX-5422 — Capsule dosed every other day for 21 days out of 28 day cycle. Dose escalation based on safety

SUMMARY:
Hsp90 is a chemical in the body that is involved int he promotion of cancer. SNX-5422 is an experimental drug that blocks Hsp90.

DETAILED DESCRIPTION:
SNX-5422 is a prodrug for SNX-2112. Correlation has been observed between Hsp90 client protein level changes and functional effects in cells in in vitro studies of SNX-2112, supporting inhibition of Hsp90 as the mechanism of action for this compound. SNX-5422 has demonstrated significant antitumor activity in mouse xenograft models of human tumors, including breast (BT474, MX-1), colon (HT29), prostate (PC3), and melanoma (A375) with multiple oral dosing regimens. Pharmacokinetic (PK) studies in mice, rats, and dogs have shown high bioavailability of SNX-2112 following oral administration of SNX 5422. In mouse xenograft studies, SNX-2112 was selectively retained in tumor tissue compared with other tissues. This study will employ critical risk management features including the use of the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, which provides a scale for consistently grading the severity of AEs, toxicity criteria analyses for dose escalation, frequent laboratory and clinical observations, correlation of AEs with plasma concentrations of SNX-5422 and SNX-2112, monitoring of the QTc interval at appropriate time points, and a conservative dose-escalation scheme.

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant, non-breastfeeding females 18 years-of-age or older with histologically confirmed non-Hodgkins lymphoma, without known or clinically suspected CNS involvement, that is refractory to available therapy or for which there is no available therapy.
* No more than 4 prior lines of systemic anti-cancer therapy and no prior bone marrow transplant or stem cell transplant within 12 months of dosing, and no prior allogeneic transplant.
* Karnofsky performance score ≥60
* Life expectancy of at least 3 months.
* Adequate baseline laboratory assessments

Exclusion Criteria:

* Currently receiving anticancer therapy or have received anticancer therapy within the past 28 days or 5 half-lives of the anticancer therapy
* The need for treatment with medications with clinically-relevant metabolism by the cytochrome P450 (CYP) 3A4 isoenzyme within 3 hours before or after administration of SNX-5422
* At increased risk for developing prolonged QT interval, including hypokalemia or hypomagnesemia, unless corrected to within normal limits prior to first dose of SNX-• Chronic diarrhea.
* Gastrointestinal diseases or conditions that could affect drug absorption, including gastric bypass.
* Gastrointestinal diseases that could alter the assessment of safety, including irritable bowel syndrome, ulcerative colitis, Crohn's disease, or hemorrhagic coloproctitis.
* History of documented adrenal dysfunction not due to malignancy.
* Seropositive for human immunodeficiency virus (HIV) or hepatitis C virus (HCV).
* History of chronic liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Number of patients with dose limiting toxicities | First 28 day cycle
  Number of patients with dose-limiting toxicities defined as AEs or laboratory abnormalities of Common Terminology Criteria for Adverse Events [CTCAE] version 4.03 ≥ Grade 3 that are not clearly related to disease progression

SECONDARY OUTCOMES:
Number of patients with adverse events as a measure of tolerability | Day 28 of each cycle
  Frequency and severity of AEs, changes in vital signs, ECG, physical examination and clinical chemistry, hematology and urinalysis
Tumor progression | Completion of every two 28 day cycles
  Hematological disease assessment of all known sites of disease using the appropriate hematological malignancy response criteria compared to baseline

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - Georgia Regents University Cancer Center, Augusta, Georgia
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee